CLINICAL TRIAL: NCT02500069
Title: The Effect of Intestinal Brake Activation at Different Locations in the Gut on Food Intake and Hormone Release
Brief Title: Location Specific Differences in Intestinal Brake Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: METC-14-3-006
Record Dates: First submitted 2014-03-18; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Ileal Brake; Satiety; Overweight; Obesity; Overeating
MeSH Terms: conditions — Overweight; Obesity; Hyperphagia | interventions — Caseins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Tap water infusion in all three locations (duodenum, jejunum and ileum)
  Interventions: Other: placebo
- Duodenum (Experimental): Infusion of casein in duodenum
  Interventions: Other: Casein (in duodenum)
- Jejunum (Experimental): Infusion of casein in jejunum
  Interventions: Other: Casein (in jejunum)
- Ileum (Experimental): Infusion of casein in ileum
  Interventions: Other: Casein (in ileum)

INTERVENTIONS:
Other: placebo — infusion of tap water in all regions (duodenum, jejunum and ileum)
  Arms: Placebo
Other: Casein (in duodenum) — infusion of protein in duodenum
  Arms: Duodenum
Other: Casein (in jejunum) — infusion of protein in jejunum
  Arms: Jejunum
Other: Casein (in ileum) — infusion of protein in ileum
  Arms: Ileum

SUMMARY:
The appearance of intact macronutrients in the small intestine can result in the activation of an intestinal brake; a negative feedback mechanism from different parts of the intestine to the stomach, the small intestine and to the central nervous system. These processes inhibit food processing, appetite sensations and food intake, and furthermore they increase feelings of satiety and satiation. The researchers will investigate the effects of intraduodenal, intrajejunal and intralileal infusion of casein (protein) on ad libitum food intake, satiation and in vivo release of the gut satiety peptides CCK, PYY and GLP-1 and glucose and insulin.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Based on medical history and previous examination, no gastrointestinal complaints can be defined.
* Age between 18 and 65 years. This study will include healthy adult subjects (male and female). Women must be taking contraceptives.
* BMI between 18 and 25 kg/m2)
* Weight stable over at least the last 6 months (≤5% weight change)

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
* Use of medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator)
* Dieting (medically prescribed, vegetarian, diabetic, macrobiological, biological dynamic)
* Pregnancy, lactation
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* Smoking
* Blood donation within 3 months before the study period
* Self-admitted HIV-positive state
* Weight <60kg
* Evidence of casein or sucrose hypersensitivity
* Participation in any other study in which radiation was used, within 12 months before the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To measure ad libitum food intake at the end of the test day | 1 test day
  Food intake measurement in kcal

SECONDARY OUTCOMES:
VAS scores for hunger and satiety | 1 test day
  Visual analogue scale for hunger and satiety in mm (0-100 mm scale)
GI peptides | 1 test day
  Measurement of GI peptide release during protein infusion (CCK, GLP-1, PYY, insulin and glucose)

CONTACTS AND LOCATIONS:
Overall Officials: A Masclee, Prof. dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] van Avesaat M, Ripken D, Hendriks HF, Masclee AA, Troost FJ. Small intestinal protein infusion in humans: evidence for a location-specific gradient in intestinal feedback on food intake and GI peptide release. Int J Obes (Lond). 2017 Feb;41(2):217-224. doi: 10.1038/ijo.2016.196. Epub 2016 Nov 4. PMID 27811949